CLINICAL TRIAL: NCT01349257
Title: Study Title: A Single-dose, Open-label, Randomised, 2-way Crossover, Clinical Pharmacology Study of Four Inhalations of CHF 1535 100/6 NEXT DPI® (Fixed Combination of Beclomethasone Diproponate 100 µg Plus Formoterol Fumarate 6 µg) Versus the Same Dose of CHF 1535 100/6 pMDI Both Administered With Charcoal Block.
Brief Title: Pharmacokinetic Clinical Study of CHF1535 NEXT DPI® Versus CHF1535 pMDI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCD-1015-PR-0055; 2010-024384-40 (EudraCT Number)
Record Dates: First submitted 2011-04-22; First posted 2011-05-06 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Asthma
Keywords: Asthmatic patients
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: BDP/Formoterol — One single day treatment of CHF 1535 100/6 NEXT DPI®: CHF 1535 dry powder for inhalation (fixed combination of beclomethasone dipropionate 100 µg plus formoterol fumarate 6 µg per actuation) administered via the NEXT DPI® dry powder inhaler with charcoal block.

SUMMARY:
The aim of this clinical study is to compare the lung exposure of the contents of the trial drug after administration of the fixed combination between beclomethasone and formoterol delivered via the new Chiesi dry powder inhaler in comparison to the beclomethasone and formoterol delivered via the pressurised metered dose inhaler (pMDI) using a spacer device. To determine lung exposure, the treatments are administered with charcoal block.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults (≥18 and ≤ 70 years old).
2. Written informed consent obtained by the patient prior to any study-related procedures.
3. Diagnosis of asthma as defined by the GINA guidelines, update 2009, at least in the 6 months before the screening visit.
4. Asthmatic patients already treated with low or medium daily dose of ICS (e.g. BDP or equivalent ≤ 1000 µg/die) or low dose of ICS/LABA fixed combination (e.g. salmeterol/fluticasone 100/500 µg/die).
5. Patients with a pre-bronchodilator forced expiratory volume in one second (FEV1) ≥ 60% and ≤ 90% of the predicted values.
6. Non or ex-smokers who smoked less than 5 pack-years and stopped smoking for at least 1 year. (Pack/year: number of cigarette smoked per day multiplied by the number of years of smoking/20).
7. Ability to a proper use of pMDI plus spacer and DPI devices.
8. A cooperative attitude to be compliant with study procedures.
9. Body mass index (BMI) ≥18.5 and ≤ 32 kg/m2

Exclusion Criteria:

1. Pregnant or lactating women or all women physiologically capable of becoming pregnant UNLESS they meet the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea or are using one or more of the following acceptable methods of contraception.

   * surgical sterilization (e.g. bilateral tubal ligation, hysterectomy)
   * hormonal contraception (implantable, patch, oral)
   * other forms of effective contraception including placement of an intrauterine device (IUD) or intrauterine system (IUS) or barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal cream/foam/gel/ suppository.
2. Significant seasonal variation in asthma or asthma occurring only during episodic exposure to an allergen or a chemical sensitizer.
3. History of near fatal asthma (e.g. brittle asthma, hospitalization for asthma exacerbation in Intensive Care Unit).
4. Patients with abnormal QTcF at Screening Visit: QTcF > 450 msec for male subjects and QTcF > 470 msec for female subjects.
5. Diagnosis of COPD as defined by the current GOLD guidelines, updates 2009.
6. Hospitalization due to asthma exacerbation within 1 month prior to the screening visit or during the run-in period.
7. Lower respiratory tract infection within one month prior to screening until randomization.
8. History of cystic fibrosis, bronchiectasis or alpha-1 antitrypsin deficiency.
9. History of drug addiction or excessive use of alcohol (weekly intake in excess of 28 units alcohol; one unit being a glass of beer, wine or a measure of spirits), or excessive consumption of xanthine containing substances (daily intake in excess of 5 cups of coffee, tea, cola, etc) or psychological or other emotional problems likely to invalidate informed consent, or limit the ability of the subject to comply with the protocol requirements;
10. Diagnosis of restrictive lung disease.
11. Patients treated with oral or parenteral corticosteroids in the previous 2 months before the screening visit (3 months for parenteral depot corticosteroids).
12. Intolerance or contra-indication to treatment with beta2-agonists and/or inhaled corticosteroids or allergy to any component of the study treatments.
13. Having received an investigational drug within 1 month before the screening visit.
14. Significant medical history of and/or treatments for cardiac, renal, neurological, hepatic, endocrine diseases, or any laboratory abnormality indicative of a significant underlying condition, that may interfere with patient's safety, compliance, or study evaluations, according to the investigator's opinion.
15. Any patient with active cancer or a history of cancer with less than 5 years disease free survival time (whether or not there is evidence of local recurrence or metastases). Localized basal cell carcinoma (without metastases) of the skin is acceptable.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
lung bioavailability | 13 times/24hr
  To compare the lung bioavailability of B17MP (active metabolite of BDP) and formoterol after four inhalations using the new Chiesi dry powder inhaler vs pMDI using spacer device, with activated Charcoal Block.

SECONDARY OUTCOMES:
To assess the safety and the tolerability of the study treatments considering AE and measuring vitals signs as blood pressure and heart rate in the specified time frame. | 13 times/24hr
  Adverse events and Vital signs: blood pressure and heart rate assessed at pre-dose and 30 min, 1, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Principal Investigator — Medicines Evaluation Unit Ltd, Manchester, United Kingdom
Locations (1):
- Medicines Evaluation Unit Ltd, Manchester, United Kingdom

REFERENCES:
- [Result] Govoni M, Piccinno A, Lucci G, Poli G, Acerbi D, Baronio R, Singh D, Kuna P, Chawes BL, Bisgaard H. The systemic exposure to inhaled beclometasone/formoterol pMDI with valved holding chamber is independent of age and body size. Pulm Pharmacol Ther. 2015 Feb;30:102-9. doi: 10.1016/j.pupt.2014.04.003. Epub 2014 Apr 16. PMID 24746942
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2010-024384-40